CLINICAL TRIAL: NCT04534764
Title: Evaluation of Visual Performance of Two Types of Cosmetic Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-6060
Record Dates: First submitted 2020-08-11; First posted 2020-09-01 (Actual); Results first posted 2021-09-01 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- TEST/CONTROL (Experimental): Eligible subjects that are habitual soft contact lens wearers will be randomized into lens wear sequence (Test/Control)
  Interventions: Device: etafilcon A with cosmetic pattern; Device: 1-Day Acuvue DEFINE Vivid Style
- CONTROL/TEST (Experimental): Eligible subjects that are habitual soft contact lens wearers will be randomized into lens wear sequence (Control/Test)
  Interventions: Device: etafilcon A with cosmetic pattern; Device: 1-Day Acuvue DEFINE Vivid Style

INTERVENTIONS:
Device: etafilcon A with cosmetic pattern — TEST
Device: 1-Day Acuvue DEFINE Vivid Style — CONTROL

SUMMARY:
This is a single visit, brand-masked, non-dispensing, 2×2 bilateral crossover study. Each subject will be bilaterally fitted with one of the two test articles in each of the study periods in a random order with a 5-minute washout period in between study lenses.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled in the study:

  1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form
  2. Appear able and willing to adhere to the instructions set forth in this clinical Protocol.
  3. Subjects between 18 and 39 (inclusive) years of age at the time of screening
  4. Be a current soft contact lens wearer in both eyes with a minimum of 6 hours/day and 5 days/week over the last month by self-report.
  5. The subject must be willing to be photographed and/or video-taped.
  6. The subject's vertex corrected spherical equivalent distance refraction must be in the range of -1.00 D to -6.00 D (inclusive) in each eye
  7. The subject's refractive cylinder must be less than or equal to 0.75 D (inclusive) in each eye.
  8. Have spherical best corrected visual acuity of 20/25 or better in each eye.

     Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Currently pregnant or lactating
  2. Any systemic disease (eg, Sjögren's Syndrome), allergies, infectious disease (eg, hepatitis, tuberculosis), contagious immunosuppressive diseases (eg, HIV), autoimmune disease (eg rheumatoid arthritis), or other diseases, by self-report, which are known to interfere with contact lens wear and/or participation in the study (at the investigators discretion).
  3. Use of systemic medications (eg, chronic steroid use) that are known to interfere with contact lens wear (at the investigators discretion)
  4. Any previous, or planned (during the study) ocular surgery (eg, radial keratotomy, PRK, LASIK, etc.)
  5. Participation in any contact lens or lens care product clinical trial within seven (7) days prior to study enrollment
  6. Employee or family members of clinical site (eg, Investigator, Coordinator, Technician).
  7. Any ocular allergies, infections or other ocular abnormalities that are known to interfere with contact lens wear and/or participation in the study. This may include, but not be limited to entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or corneal distortion (at the investigators discretion).
  8. Clinically significant (Grade 3 or 4 on FDA scale) tarsal abnormalities, bulbar injection, corneal edema, corneal vascularization, corneal staining, or any other abnormalities of the cornea which would contraindicate contact lens wear.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2020-08-12 (Actual); Study Completion 2020-08-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Maitland Vision Center, Maitland, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 35 subjects were enrolled in this study. Of those enrolled, all 35 subjects were dispensed both study lenses and completed the study.
Groups:
- Test/Control: Subjects randomized to receive the Test lens during the first period and then received the Control lens during the second period.
- Control/Test: Subjects randomized to receive the Control lens during the first period and then received the Test lens during the second period.
Period: Period 1
Arm/Group | Test/Control | Control/Test
Started | 18 | 17
Completed | 18 | 17
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Test/Control | Control/Test
Started | 18 | 17
Completed | 18 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: All subjects who had successfully completed all visits and did not substantially deviate from the protocol.
Arm/Group | Total
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.2 (5.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 4
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1
  Black or African American | 1
  White | 32
  Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Distance Monocular Visual Acuity (logMAR)
Description: Visual acuity on logMAR (Logarithm of Minimal Angle of Resolution) scale was evaluated at distance (4 meters) under high luminance low contrast and low luminance high contrast lighting conditions using ETDRS (Early Treatment Diabetic Retinopathy Study) charts. Letter-by letter results calculated the visual performance score for each chart read. logMAR scores closer to zero, or below zero, indicate a better visual acuity. A logMAR visual performance score of 0.0 is equivalent to Snellen visual acuity of 20/20.
Time Frame: 5 min post lens insertion
Population: All subjects who had successfully completed all visits and did not substantially deviate from the protocol.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Groups:
- Test: Subjects that wore the Test lens in either the first or second period of the study.
- Control: Subjects that wore the Control lens in either the first or second period of the study.
Arm/Group | Test | Control
Number analyzed (Participants) | 35 | 35
Number analyzed (Eyes) | 70 | 70
logMAR
  High Luminance Low Contrast | -0.016 (0.1083) | -0.001 (0.1046)
  High Luminance High Contrast | -0.171 (0.0857) | -0.151 (0.0852)
  Low Luminance High Contrast | 0.016 (0.1008) | 0.007 (0.0814)
Statistical Analysis 1: Comparison: Test vs Control; High Luminance Low Contrast; Test type: Non-Inferiority — The non-inferiority of the Test lens relative to the Control will be concluded if the upper confidence limit of LSM difference is below the non-inferiority margin 0.05 logMAR; Mixed Models Analysis; Least Square Mean Difference = -0.016, 95% CI 2-sided [-0.039 to 0.006], Standard Error of Mean 0.0114 — LS Mean difference was calculated as Test - Control
Statistical Analysis 2: Comparison: Test vs Control; Low Luminance High Contrast; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Least Square Mean Difference = 0.009, 95% CI 2-sided [-0.014 to 0.031], Standard Error of Mean 0.0114 — LS Mean difference was calculated as Test - Control

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study. Approximately 1 day per subject.
Arm/Group | Test | Control
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-21): https://cdn.clinicaltrials.gov/large-docs/64/NCT04534764/Prot_SAP_000.pdf